CLINICAL TRIAL: NCT03723135
Title: Expanded Access for CC-486
Status: Approved for marketing | Type: Expanded Access
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-486
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Acute Myelogenous Leukemia (AML)
Keywords: Expanded Access; Compassionate Use
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — cc-486; Azacitidine

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: CC-486 — Oral azacitidine administered as directed by treating physician.
  Other Names: Oral Azacitidine

SUMMARY:
This is an expanded access program (EAP) for eligible participants designed to provide access to CC-486.

ELIGIBILITY:
Inclusion Criteria:

-Adult patients with documented acute myelogenous leukemia (AML) in their first complete remission (CR) or complete remission with incomplete blood count recovery (CRi) following induction therapy with or without consolidation treatment, who seek treatment with CC-486 as monotherapy to maintain their CR or CRi.

Exclusion Criteria:

* Patients with AML in CR/CRi who plan to proceed to or are waiting for a bone marrow transplant
* Patients who have received a bone marrow transplant for the treatment of AML
* Treatment of AML patients with relapse or refractory disease
* Pregnant or breast-feeding females
* Patient meets enrollment criteria and can participate in a disease-specific clinical trial

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Celgene, Summit, New Jersey, United States